CLINICAL TRIAL: NCT06126497
Title: An Open-Label Study Evaluating the Safety and Efficacy of Ropanicant in Participants With Moderate to Severe Major Depressive Disorder
Brief Title: Study Evaluating Safety and Efficacy of Ropanicant in MDD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP2S1911A4B2
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder
Keywords: SUVN-911; Phase-2; MDD; Depression; Open label
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ropanicant 45 mg qd (Experimental): The participant will take 1 tablet/day in the morning (for qd dosing)
  Interventions: Drug: Ropanicant
- Ropanicant 30 mg bid (Experimental): The participant will take 2 tablets/day (~12 hours apart for bid dosing).
  Interventions: Drug: Ropanicant
- Ropanicant 45 mg bid (Experimental): The participant will take 2 tablets/day (~12 hours apart for bid dosing).
  Interventions: Drug: Ropanicant

INTERVENTIONS:
Drug: Ropanicant — Tablet
  Other Names: SUVN-911

SUMMARY:
This is an open-label, parallel-group study to evaluate the safety and efficacy of ropanicant in participants with moderate to severe Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
Approximately 36 participants will be randomly assigned to receive ropanicant either 45 mg qd, 30 mg bid, or 45 mg bid for 2 weeks, in a ratio of 1:1:1 (12 participants in each treatment group). Following a screening period of up to 4 weeks, the participants will be treated for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the DSM-5 criteria for MDD without psychotic features and diagnosis confirmed by the Mini-International Neuropsychiatric Interview (MINI).
* Participants with a current major depressive episode of at least 4 weeks of duration prior to the screening visit.
* Participants must have an MADRS score of ≥25 at the screening and the baseline visits.
* Participants must have a score of ≥4 on Clinical Global Impression - Severity (CGI-S) Scale at the screening and the baseline visits.

Exclusion Criteria:

* Participants who meet criteria for treatment-resistant depression during the current major depressive episode, which will be defined as being non-responders (less than 50% of symptom improvement) to 2 or more depression treatment periods of adequate dose and duration as defined by the Massachusetts General Hospital (MGH) Antidepressant Treatment Response Questionnaire (ATRQ).
* Participants taking antidepressant treatment (SSRIs and SNRIs) or any medication that is contraindicated with the use of monoamine oxidase inhibitors (eg, opioids, stimulants) within 2 weeks (or 5 half-lives, whichever is longer) prior to baseline and until the end of study visit.
* Participants who do not agree to avoid tyramine rich diet from the start of dosing and until 2 weeks following last study drug administration.
* Participants who are habitual smokers or using nicotine products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From Screening to Day 21
  Frequency and severity of adverse events, treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) score. | From Baseline to Day 14
  Change from the baseline to the MADRS total score. The MADRS is a clinician-rated scale to assess depressive symptoms which consists from 10 items. The time frame for this scale is the past 7 days. Each item is scored on 7-point scale (0 [absence of symptoms] to 6 [severe]). The total score is the sum of 10 items and can take range from 0 to 60. A higher score represents a higher severity of the level of depression.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Clinical Innovations, Inc, Bellflower, California
  - NRC Research Institute, Orange, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - CenExel iResearch, LLC, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Precise Research Centers, Flowood, Mississippi
  - Neuro behavioral Clinical Research, Inc, North Canton, Ohio
  - Cedar Clinical Research, Inc., Murray, Utah
  - Eastside Therapeutic Resource, Inc. dba Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: No